CLINICAL TRIAL: NCT01472380
Title: An Open-label, Drug Interaction Study to Investigate the Effects of Steady-State Fenofibric Acid on the Single-Dose Pharmacokinetics of Efavirenz in Healthy Subjects
Brief Title: A Drug-Drug Interaction Study Between Fenofibric Acid and Efavirenz
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-028-11-1001
Record Dates: First submitted 2011-11-11; First posted 2011-11-16 (Estimated); Results first posted 2012-07-23 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
MeSH Terms: interventions — efavirenz; fenofibric acid; Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Efavirenz 600mg alone (Active Comparator): efavirenz 600mg by mouth taken on Day 1
  Interventions: Drug: efavirenz
- Efavirenz co-administered with fenofibric acid (Active Comparator): co-administered oral doses of efavirenz 600 mg and fenofibric acid 105 mg taken on Day 31
  Interventions: Drug: efavirenz; Drug: fenofibric acid 105 mg

INTERVENTIONS:
Drug: efavirenz — 600 mg
  Other Names: SUSTIVA
Drug: fenofibric acid 105 mg — fenofibric acid 105 mg
  Other Names: FIBRICOR
  Arms: Efavirenz co-administered with fenofibric acid

SUMMARY:
Efavirenz is predominantly metabolized by cytochrome P450 (CYP) 2B6. Fenofibric Acid is an inhibitor of CYP2B6. This study will evaluate the effect of multiple doses of fenofibric acid at steady-state on the pharmacokinetics of single-dose efavirenz in healthy adult subjects.

DETAILED DESCRIPTION:
Efavirenz is predominantly metabolized by cytochrome P450 (CYP) 2B6. Fenofibric Acid is an inhibitor of CYP2B6. This study will evaluate the effect of multiple doses of fenofibric acid at steady-state on the pharmacokinetics of single-dose efavirenz in healthy adult subjects. This study will not evaluate the the effects of efavirenz on fenofibric acid pharmacokinetics. On study Day 1 after a fast of at least 10 hours, thirty healthy, non-smoking, non-obese, non-pregnant adult volunteers between the ages of 18 and 45 will be given one oral dose of efavirenz (1 x 600 mg tablet). Fasting will continue for 4 hours after the dose. Blood samples will be drawn from all participants before dosing and for 24 hours post-dose on a confined basis at times sufficient to adequately define the pharmacokinetics of efavirenz. Blood sampling will then continue on a non-confined basis at 48, 72, 96 and 120 hours post-dose. A 21 day washout period will be completed after the first dose of efavirenz on Day 1. On Days 22 through 30, all subjects will receive a single oral dose of fenofibric acid (1 x 105 mg tablet) in the morning without regard to meals. On the morning of Day 31 after a fast of at least 10 hours, all study participants will receive co-administered single oral doses of efavirenz (1 x 600 mg tablet) and fenofibric acid (1 x 105 mg tablet). Fasting will continue for 4 hours after the dose. Blood samples will be drawn from all participants before dosing and for 24 hours post-dose on a confined basis at times sufficient to adequately determine the pharmacokinetics of efavirenz. Blood sampling will then continue on a non-confined basis at 48, 72, 96 and 120 hours post-dose. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout participation in the study for adverse reactions to the study drug and/or procedures. Vital signs (seated blood pressure and pulse) will be measured prior to dosing and at approximately 1, 2, 3 and 5 hours post-dose on Days 1, 22 and 31 to coincide with peak plasma concentrations of both efavirenz and fenofibric acid. Blood pressure and pulse will also be obtained at 24 hours post-dose on Days 2 and 32 prior to discharge from the clinical study unit. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the Investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-45 years of age, non-smoking and non-pregnant (post-menopausal, surgically sterile or using effective contraceptive measures), with a body mass index (BMI) greater or equal to 18 and less than or equal to 32kg/m2, hemoglobin >12 g/dL.

Exclusion Criteria:

* recent participation (within past month) in other research studies
* Recent significant blood donation or plasma donation
* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Recent (2-year) history or evidence of alcoholism or drug abuse
* History or presence of significant cardiovascular, pulmonary, hepatic, gallbladder or biliary tract, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychiatric disease or active sexually transmitted disease
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 28 days prior to the first dose and throughout the study
* Drug allergies or sensitivities to efavirenz, fenofibrate, fenofibric acid or any component of the two formulations
* Subjects who have had a tattoo or body piercing within 30 days prior to administration of study medication

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Davis, MD, Study Chair — Mutual Pharmaceutical Company, Inc.
Locations (1):
- INC Research, Morgantown, West Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty (30) healthy, non-smoking adult male and female volunteers from the community at-large were enrolled
Groups:
- Efavirenz Alone, FFA Alone, Enfavirenz and FFA Together: On the morning of Day 1, subjects received a single dose of efavirenz 600 mg after an overnight fast of at least 10 hours, followed by a 21 day washout period. On the mornings of Days 22-30, subjects received a dose of fenofibric acid 105 mg without regard to meals. On the morning of Day 31, subjects received a co-administered single oral dose of efavirenz 600 mg and fenofibric acid 105 mg following an overnight fast of at least 10 hours
Period: Efavirenz Alone
Arm/Group | Efavirenz Alone, FFA Alone, Enfavirenz and FFA Together
Started | 30
Completed | 29
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Fenofibric Acid (FFA) Alone
Arm/Group | Efavirenz Alone, FFA Alone, Enfavirenz and FFA Together
Started | 29
Completed | 29
Not Completed | 0
Period: 1 Day Period Between Dosing
Arm/Group | Efavirenz Alone, FFA Alone, Enfavirenz and FFA Together
Started | 29
Completed | 28
Not Completed | 1
Not completed — Protocol Violation | 1
Period: Efavirenz and FFA
Arm/Group | Efavirenz Alone, FFA Alone, Enfavirenz and FFA Together
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Efavirenz Alone, FFA Alone, Enfavirenz and FFA Together
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 26.8 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 24
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that the drug reaches in the plasma for efavirenz
Time Frame: serial pharmacokinetic blood samples drawn immediately prior to dosing on Days 1 and 31 and then 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24, 48, 72, 96, and 120 hours after dose administration
Population: 28 of 30 subjects completed the entire study and had sufficient data to calculate at minimum the maximum concentration (Cmax)for efavirenz.
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- Efavirenz Alone: On the morning of Day 1, subjects received a single dose of efavirenz 600 mg after an overnight fast of at least 10 hours, followed by a 21 day washout period
- Efavirenz With Fenofibric Acid: On the morning of Day 31, subjects received a co-administered single oral dose of efavirenz 600 mg and fenofibric acid 105 mg after an overnight fast.
Arm/Group | Efavirenz Alone | Efavirenz With Fenofibric Acid
Number analyzed (Participants) | 28 | 28
ug/mL | 2.62 (0.57) | 2.63 (0.55)

2. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Time 0 to Time t[AUC(0-t)]
Description: The area under the plasma concentration versus time curve from time 0 to the time of the last measurable concentration (t), as calculated by the linear trapezoidal rule for efavirenz
Time Frame: as for outcome 1
Population: 28 of 30 subjects completed the entire study and had sufficient data to calculate at minimum the area under the plasma concentration versus time curve from time 0 to the time t of the last quantifiable concentration (AUC0-t) for efavirenz.
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | Efavirenz Alone | Efavirenz With Fenofibric Acid
Number analyzed (Participants) | 28 | 28
h*ug/mL | 70.58 (17.28) | 64.62 (15.22)

3. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-infinity]
Description: The area under the plasma concentration versus time curve from time 0 to infinity. [AUC(0 to infinity)] was calculated as the sum of AUC (0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant for efavirenz.
Time Frame: serial pharmacokinetic blood samples drawn immediately prior to dosing on Days 1 and 31 and then 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24, 48, 72, 96, and 120 hours after dose administration
Population: 28 of 30 subjects completed the entire study and had sufficient data to calculate at minimum the area under the plasma concentration versus time curve from time 0 to infinity for efavirenz.
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | Efavirenz Alone | Efavirenz With Fenofibric Acid
Number analyzed (Participants) | 28 | 28
h*ug/mL | 121 (33.6) | 112 (30.3)

ADVERSE EVENTS:
Groups:
- Fenofibric Acid Alone: On the mornings of Days 22-30, subjects received a dose of fenofibric acid 105 mg without regard to meals.
Arm/Group | Efavirenz Alone | Fenofibric Acid Alone | Efavirenz With Fenofibric Acid
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 19/30 | 2/29 | 15/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efavirenz Alone (N=30) | Fenofibric Acid Alone (N=29) | Efavirenz With Fenofibric Acid (N=28)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 15 (17) | 0 (0) | 8 (8)
Headache (Nervous system disorders) | 6 (6) | 2 (2) | 6 (6)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Euphoric Mood (Psychiatric disorders) | 0 (0) | 0 (0) | 5 (5)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days